CLINICAL TRIAL: NCT03755115
Title: Clinical Study of PD-1 Monoclonal Antibody SHR-1210 Combined With Epirubicin in the Treatment of Extensive Small Cell Lung Cancer After First-line Treatment Failure
Brief Title: SHR-1210 Combined With Epirubicin in the Treatment of Extensive Disease Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-EPI-II
Record Dates: First submitted 2018-11-17; First posted 2018-11-27 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-11

CONDITIONS: Small Cell Lung Cancer Extensive Stage
Keywords: ICD; PD1; ED-SCLC
MeSH Terms: interventions — Epirubicin; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epirubicin plus SHR1210 (Experimental): First intravenous injection of epirubicin injection, D1,30mg/m^2 Then intravenous administration with SHR-1210,D1, a fixed dose of 200mg, D1,30min per infusion, Q2W. The total dose of epirubicin is 360 mg/m^2.next SHR-1210 single drug maintenance .Until to secdonary disease progression or intolerance side effects.Evaluate efficacy every 3 cycles.
  Interventions: Drug: Epirubicin plus SHR1210

INTERVENTIONS:
Drug: Epirubicin plus SHR1210 — First intravenous injection of epirubicin injection, D1,30mg/m^2 Then intravenous administration with SHR-1210,D1, a fixed dose of 200mg, 30min per infusion, Q2W. The total dose of epirubicin is 360 mg/m^2.next SHR-1210 single drug maintenance .Until to secdonary disease progression or intolerance side effects.Evaluate efficacy every 3 cycles.

SUMMARY:
Patients with extensive disease SCLC after failure of first-line treatment were enrolled with SHR-1210 and epirubicin for 3 cycles to evaluate initial efficacy

DETAILED DESCRIPTION:
Small cell lung cancer is a neuroendocrine tumor with strong invasiveness, rapid growth rate and early metastasis in lung cancer. The systemic chemotherapy response rate is high in a wide range of patients, but it is easy to resist drug recurrence, which brings certain difficulties to clinical treatment. The signaling pathway activated by programmed cell death receptor 1 (PD-1) and its ligand (programmed death-ligand 1, PDL1) is a hotspot in recent years and has brought good news to cancer patients. However, PD1 inhibitors are only about 13% effective in treating lung cancer patients. Epirubicin is a classic drug that activates the immunogenicity of tumor tissues, induces tumor immunogenic death, and releases some marker proteins such as CRT, HMGB1, HSP and so on. These two drugs combine to enhance the anti-tumor effect of the human immune system.The investigators designed the study to explore the possibility of apatinib as the Second-line Therapy in ED-SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is 18-75 years old when the informed consent form is signed, and the gender is not limited.
2. Histological or cytological diagnosis of patients with extensive small cell lung cancer (ED-SCLC).
3. Must provide specimens of tumor tissue at or after diagnosis of advanced or metastatic tumors or consent to biopsy, formalized or freshly obtained, formalin-fixed, paraffin-embedded (FFPE) within 1 month prior to the first dose. After the tumor tissue block can cut at least 10 slices for staining and detection.
4. Subjects have undergone rapid progression or relapse of drug resistance after first-line treatment.
5. According to the RECIST 1.1 standard, subjects must have a target lesion that can be measured by CT or MRI.

6, ECOG PS score: 0-1 points. 7. The expected survival period is ≥ 3 months. 8, the main organ function meets the following criteria: a) blood routine (no blood transfusion within 14 days, no G-CSF, no use of drugs to correct): absolute neutrophil ≥ 1.5 × 109 / L, platelets ≥ 100 × 109 / L, hemoglobin ≥ 90 g / L, white blood cells ≥ 4.0 × 109 / L and ≤ 15 × 109 / L; b) blood biochemistry: total bilirubin ≤ 1.5 ULN, AST / ALT ≤ 2.5 ULN, (if liver metastasis, then ≤ 5 times the upper limit of normal value), ALB ≥ 30 g / L, serum creatinine ≤ 1.5 ULN; c) Coagulation function: APTT ≤ 1.5 × ULN and prothrombin time - international normalized ratio (PT-INR) < 1.5xULN ( Did not receive anticoagulant therapy).

9. Volunteer to participate in clinical trials and sign informed consent, good compliance

Exclusion Criteria:

1. Target disease exclusion criteria: 1) Exclude subjects without measurable lesions 2) Subjects who can be surgically resected or radically treated. 3) Subjects who have received anti-PD-1 (L1) or CTLA4 mAb treatment.

History and comorbidities: 1) Exclude any active, known or suspected autoimmune disease in the subject 2) Exclude 2, use anti-tumor vaccine or other anti-tumor with immune stimulation within 1 month before the first dose Subjects treated with drugs. 3) Exclude subjects who are highly suspected of having interstitial pneumonia. 4) Subjects who excluded other active malignancies requiring simultaneous treatment excluded subjects with grade II or higher myocardial ischemia or myocardial infarction, poorly controlled arrhythmias, and grade III to IV cardiac insufficiency. 5) Exclude subjects with active tuberculosis (TB). 6) Exclude subjects who had severe infections within 4 weeks prior to the first dose. Exclude subjects with any active infection. 7) Exclude subjects who are ready or have undergone tissue/organ transplantation. 8) Exclude subjects who have been vaccinated or will be vaccinated within 30 days prior to the first dose.

3. Physical examination and laboratory examinations 1) A known history of human immunodeficiency virus (HIV) is known or known to have acquired immunodeficiency syndrome (AIDS). 2) Untreated active hepatitis. 3) Exclude subjects with uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.

4, allergic reactions and adverse drug reactions 1) severe allergic reactions to other monoclonal antibodies. 2) Allergic or intolerant to the infusion. 3) Serious intolerance to epirubicin or toxicity.

5. Exclude subjects with mental illness, alcoholism, refrain from quitting, drug use or substance abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-10-28 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 month
  Objective Response Rate

SECONDARY OUTCOMES:
PFS | 2 years
  Progression Free Survival
DCR | 2 years
  Disease Control Rate
OS | 2 years
  Overall Survival
AE | 2 year
  Adverse reactions
characteristic antigen on the surface of immunogenic dead cells | 3 month
  characteristic antigen on the surface of immunogenic dead cells,such as CRT(calnetulin),HSP(heat shock protein),HMGB1(High-mobility group box 1 protein),TIL (tumor infiltrating lymphocytes)，ATP,which are measured by IHC or ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Tongde Tian, Principal Investigator — Henan Cancer Hospital (The Affiliated Cancer Hospital of Zhengzhou University)
Locations (1):
- Tian Tongde, Zhengzhou, Henan, China